CLINICAL TRIAL: NCT03170037
Title: Comparison of Two-hand Mask Ventilation Technique: Standard V-E Versus Reversal V-E Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Canlas, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 170299
Record Dates: First submitted 2017-05-15; First posted 2017-05-30 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Intubation

STUDY DESIGN:
Intervention Model Description: Comparison of 2 two-handed mask ventilation techniques' ease to anesthesia providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard V-E ventilation technique (Active Comparator): After induction of anesthesia subject will be ventilated using the standard V-E ventilation technique. Ventilation will be carried out using pressure mode ventilation at respiratory rate of 10 breaths per minute, I:E ratio of 1:2, peak inspiratory pressure of 20cmH2O and no PEEP. If the subjects can be adequately ventilated, as defined by perceivable chest movement and end tidal CO2 during the first three breaths, ventilation will continue for total ten breaths.
  Interventions: Procedure: Standard V-E ventilation technique
- Reversal V-E ventilation technique (Experimental): After induction of anesthesia subject will be ventilated using the reversal V-E ventilation technique. Ventilation will be carried out using pressure mode ventilation at respiratory rate of 10 breaths per minute, I:E ratio of 1:2, peak inspiratory pressure of 20cmH2O and no PEEP. If the subjects can be adequately ventilated, as defined by perceivable chest movement and end tidal CO2 during the first three breaths, ventilation will continue for total ten breaths.
  Interventions: Procedure: Reversal V-E ventilation technique

INTERVENTIONS:
Procedure: Standard V-E ventilation technique — For the two-handed standard V-E technique, the facemask is first placed over the bridge of the nose and mouth and then held in place by performing at two-handed jaw thrust maneuver with the index and second finger of each hand and maintaining mask contact with the patient's face by using both thumbs with mouth open. A head-tilt is performed by applying a caudal force on the mandible and mask.
  Arms: Standard V-E ventilation technique
Procedure: Reversal V-E ventilation technique — While using reversal V-E technique, the anesthesia provider stands 180 degrees opposite from the head of the bed. Thenar eminence and thumbs secure the mask around the nose while the remaining fingers pull the mandible anteriorly while keeping the mouth open.
  Arms: Reversal V-E ventilation technique

SUMMARY:
This study hypothesizes that a novel reversal V-E ventilation technique will retain its high efficiency as that of standard V-E technique and will be easier to use.

DETAILED DESCRIPTION:
Despite advances in intubation technology, difficult airways persist. Because it is failure to oxygenate, not failure to intubate, that ultimately leads to brain injury and cardiovascular collapse, effective mask ventilation is at least as important as successful intubation. Therefore optimizing mask ventilation is crucial for clinicians. When difficult mask ventilation encounters, clinicians often switch to two hand technique to hold the mask including either "C-E" clamp or "V-E" clamp. Both volume mode ventilation and pressure mode ventilation are superior with the V-E technique as compared to the C-E technique. The study will test the hypothesis that a novel reversal V-E mask ventilation technique will retain its high efficiency as that of standard V-E technique but be easier to use than standard V-E technique.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Requiring general anesthesia
* BMI =>30

Exclusion Criteria:

* Untreated ischemic heart diseases
* Respiratory disorders, including COPD and asthma
* American Society of Anesthesiologists(ASA) physical class of 4 or greater
* Undergoing emergency surgery
* Requiring rapid sequence intubation for aspiration protection
* Non propofol - induction of anesthesia
* Requiring fiberoptic intubation
* Pregnant women or women who have given birth within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Visual score of friendliness of mask holding technique using 11 point scale | Conclusion of masked ventilation (approximately 5 minutes)
  Visual score of friendliness of mask holding technique using 11 point scale when 0 is easy and 10 is difficult.

SECONDARY OUTCOMES:
AUC of exhaled tidal volume (Vt) trace | Period of masked ventilation (approximately 5 minutes)
  Comparison of AUC of exhaled tidal volume trace
Vt/AUC | Period of masked ventilation (approximately 5 minutes)
  Vt/AUC of exhaled Vt
Peak inspiratory airway pressure | Period of masked ventilation (approximately 5 minutes)
  Peak inspiratory airway pressure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Canlas, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No